CLINICAL TRIAL: NCT06871449
Title: Investigation Of The Effects Of Unilateral And Bilateral Spinal Anesthesia On Cerebral Blood Flow
Status: Completed | Type: Observational
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, MEHTAP BALCI, Assistant Professor, Nuh Naci Yazgan University
Other Study IDs: Mehtap Balcı
Record Dates: First submitted 2025-01-19; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Adverse Effect; Cerebral Perfusion
Keywords: Spinal Block, Near-Infrared Spectroscopy ,Cerebral Oxygenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unilateral Spinal Block(GroupI): Group I: After appropriate area cleaning, under sterile conditions, the spinal space was accessed through the L4-L5 interspace, and 15 mg of hyperbaric bupivacaine (3 cc, Buvasin 0.5% Spinal Heavy) was administered following the observation of free, clear cerebrospinal fluid (CSF) flow. The patient was then kept in the lateral position on the surgical side for 5 minutes before being moved to the supine position.
- Bilateral Spinal Block (Group II): Group II: After appropriate area cleaning, under sterile conditions, the spinal space was accessed through the L4-L5 interspace, and 15 mg of hyperbaric bupivacaine (3 cc, Buvasin 0.5% Spinal Heavy) was administered following the observation of free, clear cerebrospinal fluid (CSF) flow. The patient was then kept in the supine position for 5 minutes.

SUMMARY:
Spinal anesthesia is a widely used method in anesthesia practice. Unilateral spinal block refers to a neuroaxial technique that induces motor and sensory blockade on the surgical side. While spinal anesthesia offers numerous advantages, it is associated with complications such as hypotension, headache, transient neurological symptoms, and meningitis. Among these, hypotension is the most common. To mitigate hemodynamic issues, intravenous fluid preloading and vasopressor use are standard practices in many centers.

This study aimed to compare regional cerebral oxygenation (rSO₂) values in patients undergoing unilateral and bilateral spinal blocks to identify the least complicated and most effective method. Minimizing complications can facilitate early mobilization, reduce hospital stays, and lower infection risks.

The study included 60 male patients (aged 18-65 years) scheduled for unilateral inguinal hernia surgery at Kayseri City Hospital. Inclusion criteria were the absence of coagulation disorders, infections, or systemic diseases, hemoglobin levels >10 g/dL, and BMI <30. Patients were randomized into two groups:

Group I: Unilateral spinal anesthesia with 15 mg hyperbaric bupivacaine. Patients were placed in a lateral position on the surgical side for 5 minutes, then moved to the supine position.

Group II: Bilateral spinal anesthesia with 15 mg hyperbaric bupivacaine. Patients were placed in the supine position for 5 minutes.

Sensory block levels were assessed using the pin-prick test, and motor blocks were evaluated with the Bromage scale. Surgery commenced when the sensory block reached the T10 level. Patient data, including age, BMI, hemoglobin, baseline systolic/diastolic blood pressure (SBP/DBP), mean arterial pressure (MAP), heart rate (HR), oxygen saturation (SpO₂), and rSO₂, were recorded before and after spinal anesthesia. SBP, DBP, MAP, HR, SpO₂, and rSO₂ values were monitored at 5-minute intervals for 30 minutes.

DETAILED DESCRIPTION:
This study was conducted with the approval of the Kayseri City Hospital Scientific Research and Publication Ethics Committee (approval number: 2022/605). Written informed patient consent was obtained (A Guide to Good Clinical Practice, 609, Mehtap Balcı, 24.03.2022). This manuscript adheres to the applicable TITCK - Turkish Pharmaceutical and Medical Device Authority guideline. It was determined that meaningful results could be obtained with a minimum of eight patients by performing a power analysis.

A total of 60 male volunteer patients, aged 18-65 years, scheduled for unilateral inguinal hernia surgery in the Kayseri City Hospital operating room, were included. The inclusion criteria were the absence of coagulation disorders or prolonged bleeding times, no infections at the injection site or systemic infections, ability to cooperate, no history of opioid use or local anesthetic allergy, no cardiovascular, respiratory, or metabolic diseases, hemoglobin levels >10 g/dL, and BMI <30. Patients were randomly assigned to two groups of 30 each.

Before surgery, patients were informed about the procedure and the anesthesia method. After reading and signing the informed consent form, volunteer patients were brought to the operating table. Intravenous access was established for all patients, and non-invasive monitoring was initiated. Patients were placed in a seated position, and the intervention area was cleaned with 10% povidone-iodine. Under sterile conditions, a 22G (Quincke) spinal needle was slowly advanced into the L4-5 spinal interspace, and free, clear cerebrospinal fluid (CSF) flow was observed.

Group I: Spinal anesthesia was performed with 15 mg of hyperbaric bupivacaine (3 cc, Buvasin 0.5% Spinal Heavy), followed by placing the patient in a lateral position on the surgical side for 5 minutes and then switching to the supine position.

Group II: Spinal anesthesia was performed with 15 mg of hyperbaric bupivacaine (3 cc, Buvasin 0.5% Spinal Heavy), followed by placing the patient in the supine position for 5 minutes.

The sensory block level was assessed using the pin-prick test, and the motor block level was evaluated using the Bromage scale. Surgery commenced once the sensory block reached the T10 level. Throughout the surgery, all patients received 3 L/min of 100% oxygen via a face mask.

Groups:

Group I: Intrathecal 15 mg hyperbaric bupivacaine (3 cc), lateral position for 5 minutes.

Group II: Intrathecal 15 mg hyperbaric bupivacaine (3 cc), supine position for 5 minutes.

Data regarding the patients' demographic characteristics (age, height, weight, BMI), baseline hemoglobin (Hb), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), oxygen saturation (SpO₂), and regional cerebral oxygenation (rSO₂) were recorded before and after spinal anesthesia. SBP, DBP, MAP, HR, SpO₂, and rSO₂ values were recorded at 5, 10, 15, 20, 25, and 30 minutes after spinal anesthesia. The data obtained will be analyzed using SPSS 25. If the parametric assumptions (Shapiro-Wilk test) are met, a t-test will be applied to determine the significance of the difference between independent groups, and variance analysis (ANOVA) will be applied for repeated measurements within groups.

ELIGIBILITY:
Inclusion Criteria:

* No coagulation disorders or prolonged bleeding times
* No infections at the injection site or systemic infections
* Ability to cooperate
* No history of opioid use or local anesthetic allergy
* No cardiovascular, respiratory, or metabolic diseases
* Hemoglobin levels >10 g/dL
* BMI <30

Exclusion Criteria:

* Coagulation disorders present
* Infections at the injection site or systemic infections
* Inability to cooperate
* History of opioid use or local anesthetic allergy
* Cardiovascular, respiratory, or metabolic diseases present
* Hemoglobin levels <10 g/dL
* BMI >30

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 60 male volunteer patients, aged 18-65 years, scheduled for unilateral inguinal hernia surgery in the operating room of Kayseri City Hospital, were included.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Regional Cerebral Oxygenation | 5-minute intervals for 30 minutes.
  rSO₂ values were monitored

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan Üniversity Faculty of Dentistry, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kusku A, Demir G, Cukurova Z, Eren G, Hergunsel O. Monitorization of the effects of spinal anaesthesia on cerebral oxygen saturation in elder patients using near-infrared spectroscopy. Braz J Anesthesiol. 2014 Jul-Aug;64(4):241-6. doi: 10.1016/j.bjane.2013.06.012. Epub 2013 Oct 18. PMID 24998107
- [Result] Nishikawa K, Hagiwara R, Nakamura K, Ishizeki J, Kubo K, Saito S, Goto F. The effects of the extent of spinal block on the BIS score and regional cerebral oxygen saturation in elderly patients: A prospective, randomized, and double-blinded study. J Clin Monit Comput. 2007 Apr;21(2):109-14. doi: 10.1007/s10877-006-9063-7. Epub 2007 Jan 10. PMID 17216322
- [Result] Minville V, Asehnoune K, Salau S, Bourdet B, Tissot B, Lubrano V, Fourcade O. The effects of spinal anesthesia on cerebral blood flow in the very elderly. Anesth Analg. 2009 Apr;108(4):1291-4. doi: 10.1213/ane.0b013e31819b073b. PMID 19299802
- [Result] Hoppenstein D, Zohar E, Ramaty E, Shabat S, Fredman B. The effects of general vs spinal anesthesia on frontal cerebral oxygen saturation in geriatric patients undergoing emergency surgical fixation of the neck of femur. J Clin Anesth. 2005 Sep;17(6):431-8. doi: 10.1016/j.jclinane.2004.09.013. PMID 16171663
- [Result] Hino A, Ueda S, Mizukawa N, Imahori Y, Tenjin H. Effect of hemodilution on cerebral hemodynamics and oxygen metabolism. Stroke. 1992 Mar;23(3):423-6. doi: 10.1161/01.str.23.3.423. PMID 1542907
- [Result] Sun S, Liu NH, Huang SQ. Role of cerebral oxygenation for prediction of hypotension after spinal anesthesia for caesarean section. J Clin Monit Comput. 2016 Aug;30(4):417-21. doi: 10.1007/s10877-015-9733-4. Epub 2015 Jul 18. PMID 26186992
- [Result] Aydin G, Sayan CD. Is body mass index a risk factor for low cerebral oxygenation during spinal anesthesia in women undergoing cesarean section? A preliminary study. Turk J Med Sci. 2019 Jun 18;49(3):854-861. doi: 10.3906/sag-1810-208. PMID 31190520
- [Result] Hirose N, Kondo Y, Maeda T, Suzuki T, Yoshino A. Relationship between regional cerebral blood volume and oxygenation and blood pressure during spinal anesthesia in women undergoing cesarean section. J Anesth. 2016 Aug;30(4):603-9. doi: 10.1007/s00540-016-2165-6. Epub 2016 Mar 24. PMID 27011334